CLINICAL TRIAL: NCT06359912
Title: Phase I Clinical Study on the Safety and Preliminary Efficacy of Allogeneic Endothelial Progenitor Cells (EPCs) Injection in Patients With Critical Limb Ischemia
Brief Title: Safety and Preliminary Efficacy of Allogeneic Endothelial Progenitor Cells (EPCs) in Patients With Critical Limb Ischemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Allife Medical Science and Technology Co., Ltd. (Industry)
Collaborators: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNYX-EPCs-002-1
Record Dates: First submitted 2024-03-29; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Critical Limb Ischemia
Keywords: Leg Pain; Ulcer; iscemia; Peripheral Vascular Diseases
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Ulcer; Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (clinical standard treatment, EPCs) (Experimental): Patients receive clinical standard treatment and EPCs IV with a single dose
  Interventions: Drug: EPCs; Behavioral: Clinical standard treatment (CST)
- clinical standard treatment (Other): Patients receive clinical standard treatment
  Interventions: Behavioral: Clinical standard treatment (CST)

INTERVENTIONS:
Drug: EPCs — IV
  Other Names: iPSC EPCs
  Arms: Treatment (clinical standard treatment, EPCs)
Behavioral: Clinical standard treatment (CST) — Clinical standard treatment
  Other Names: CST

SUMMARY:
The purpose of this study is to determine if allogeneic Endothelial Progenitor Cells (EPCs) intravenous infusion to a subject with leg ulcer and/or gangrene due to poor blood flow will be safe and if it will relieve leg pain, increase blood flow, and/or cure the leg wound.

DETAILED DESCRIPTION:
Critical limb ischemia (CLI) is a progressive disease, which arises as a result of atherosclerosis or vasculitis in leg arteries. Prognosis of CLI is poor, and no effective treatments have been established in patients who are not eligible for the traditional revascularization therapies such as angioplasty and bypass procedures due to the inappropriate anatomy of the leg arteries or frequent reocclusion following revascularization. Therefore, it is necessary to establish novel revascularization treatment to improve prognosis of the no-option patients. The investigators will study the safety and clinical efficiency of vascular regeneration by means of transplantation of allogeneic Endothelial Progenitor Cells in patients with CLI who are not eligible for traditional revascularization treatments. The primary endpoint is the safety and tolerance identified by adverse events related with investigated drug；while the secondary endpoints are evaluation of the preliminary efficacy of EPCs.

ELIGIBILITY:
Inclusion Criteria:

* CLI patients fulfilling all the following criteria are considered suitable for inclusion in the study.

  1. Age is between 18 and 80.
  2. Diagnosis of critical limb ischemia, no surgery or interventional therapy, or poor results one month after interventional therapy (no relief of symptoms), Rutherford grade 3, grade 4 or grade 5, while meeting one of the following criteria: 1) severe intermittent claudication; 2) resting pain; 3) ABI≤ 0.60;
  3. Within the last month, Digital Subtraction Angiography (DSA), Computed Tomography Arteriography (CTA), Magnetic Resonance Angiography (MRA)，or vascular ultrasound has confirmed that one or more of the arteries (superficial femoral artery, i.e., the femoral artery below the deep femoral artery branch, the popliteal artery, and its following arteries) have a stenosis of ≥70% or occlusion;
  4. The degree of skin ulcer is determined according to Wagner, grade less than or equal to 4;
  5. Resting pain lasted for more than 2 weeks when signing the informed consent form
  6. Eligible patients of childbearing potential (both men and women) if sexually active must agree to use a reliable method of contraception with their partners
  7. The subject or agent can understand the basic requirements of the study, provide written informed consent, and follow up according to the trial requirements.

Exclusion Criteria:

* Any one of the following exclusion criteria is sufficient to disqualify a patient from the study.

  1. Subjects who have received other cell therapies previously
  2. Subjects who have received or are attending any other unlisted clinical study drug or treatment within 4 weeks prior to the first dose;
  3. Stenosis of ≥75% in the main-iliac artery;
  4. Subjects whose Feet or lower limb infections are uncontrollable, or other uncontrolled active infections;
  5. Patients with diabetic proliferating retinopathy (diabetic retinopathy grade 4 according to the International Clinical Classification Standard for diabetic retinopathy)
  6. Acute ischemic disease of the lower limb(s) occurred within the past 2 weeks;
  7. presence of uncontrolled hypertension;
  8. Any one with cerebral infarction, cerebral hemorrhage, heart failure, unstable angina pectoris, acute myocardial infarction, or severe arrhythmia before enrollment;
  9. abnormal Laboratory tests including severe liver, kidney and coagulation disorders, severe anemia etc.
  10. Patients with severe respiratory disease and other active lung infections requiring intervention that were not eligible for participation in the study
  11. Hepatitis B surface antigen positive, hepatitis C virus antibody positive, syphilis serum antibody positive or HIV antibody positive
  12. Patients with malignancy within the 5 years prior to screening (except for cured basal cell skin carcinoma, cervical carcinoma in situ, papillary thyroid carcinoma)
  13. Patients with mental illness, cognitive impairment, except those cured of depression; estimated survival of less than 12 months
  14. Congenital or acquired immunodeficiency;
  15. Subjects with Pregnant or lactating subjects
  16. Subjects with known allergy to more than 2 drugs
  17. Current or recent history of alcohol or drug abuse
  18. Patients not eligible for enrollment as comprehensively assessed by the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
adverse events | baseline to 1 year
  Incidence and severity of adverse events assessed by CTCAE V5.0

SECONDARY OUTCOMES:
Painless walking and intermittent claudication distance | month 6
  Changes from the baseline of painless walking and intermittent claudication distance by visit
Blood flow of the affected limb | month 6
  Changes from the baseline of Blood flow of the affected limb by visit
Rutherford grade | month 6
  Changes from the baseline of Rutherford grade by visit. The range of Rutherford grade is from 0 (normal) to 6 (worse).
The area of skin ulcer | month 6
  Changes from the baseline of the area of skin ulcer by visit
Vascular Quality of Life Questionnaire-6 score | month 6
  Changes from the baseline of Vascular Quality of Life Questionnaire-6 score by visit. The range of scores is from 6 (normal) to 24.

CONTACTS AND LOCATIONS:
Locations (1):
- Hui Shi, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No